CLINICAL TRIAL: NCT00329771
Title: Brush Allodynia in Patients With Episodic Migraine During an Acute Attack.
Brief Title: Research Study to Determine Sensitivity to Gentle Touch and Pressure During an Active Migraine Attack.
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: EM-BA/AAA
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Episodic migraineurs: Eligible subjects with episodic migraine (with or without aura)
  Interventions: Other: No intervention: We are testing for the presence of allodynia

INTERVENTIONS:
Other: No intervention: We are testing for the presence of allodynia — We are testing for the presence of abnormal sensation (allodynia) during a migraine attack.

SUMMARY:
Cutaneous allodynia (pronounced q-tane-ee-us all-o-din-ee-a) is common in migraine. It is a heightened skin sensitivity during an active migraine attack. Migraine attacks in patients who experience allodynia are more difficult to treat. This study intends to collect and evaluate data on the phenomenon of allodynia in patients with episodic migraine during an actual attack. The results of this study may help clinicians better understand allodynia, thereby helping them diagnose and more effectively manage patients with migraine and allodynia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65, inclusive
* Diagnosis of episodic migraine with or without aura.
* Ability to read and understand an informed consent form and study procedures

Exclusion Criteria:

* Patients with abnormal sensory findings on examination, or any known neurological disease that may affect skin sensation (peripheral neuropathy, multiple sclerosis, stroke, etc).
* Patients who suffer from headache (of any type) 15 or more days per month
* Patients who are cognitively impaired, as determined by investigator
* Patients with significant psychiatric disorder that may affect their understanding of the study protocol and/or their cooperation with the investigators.
* Patients who had taken any acute pain medication (e.g. triptans, ergots, NSAIDs, opioids, butalbital, acetaminophen) for any indication within 12 hours prior to allodynia testing.
* Patients with skin diseases that may cause abnormal skin sensation.
* Patients who had been treated with a nerve block in the 4 week period prior to allodynia testing Patients who had been treated with Botulinum neurotoxin within the 4 month period prior to allodynia testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with episodic migraine, as defined by the International Headache Society,recruited from our office practice and the communitiy
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham A Ashkenazi, M.D., Principal Investigator — Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Episodic Migraineurs
Started | 28
Completed | 25 (3 subjects withdrew or were lost to follow-up)
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Episodic Migraineurs
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Allodynia During a Migraine Attack
Description: Brush allodynia (discomfort with normal sensation) measured at pre-specified sites on the head, neck and forearms using a 100 mm visual analog scale (VAS). After each series of brushes the patient will be asked to rate the level of discomfort from "normal sensation" to "extremely painful or unpleasant" using a 100 mm visual analog scale (VAS).
Time Frame: allodynia assessed within 4 hours from onset of migraine head pain
Population: Participants who completed allodynia test
Measure: Number; unit: participants
Arm/Group | Episodic Migraineurs
Number analyzed (Participants) | 25
participants | 15

ADVERSE EVENTS:
Arm/Group | Episodic Migraineurs
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No